CLINICAL TRIAL: NCT04512716
Title: Iomab-ACT: A Pilot Study of 131-I Apamistamab Followed by CD19-Targeted CAR T-Cell Therapy for Patients With Relapsed or Refractory B-Cell Acute Lymphoblastic Leukemia or Diffuse Large B-Cell Lymphoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-382
Record Dates: First submitted 2020-07-28; First posted 2020-08-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: B-ALL; DLBCL; B ALL; Dlbcl-Ci; DLBCL Unclassifiable; DLBCL, Nos Genetic Subtypes; DLBCL Activated B-Cell Type; DLBCL Germinal Center B-Cell Type; Diffuse Large B-cell Lymphoma; HGBL; HGBL, Nos
Keywords: CD19+ B-cell malignancy; 131-I apamistamab; B-cell malignancy; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Pyloric Stenosis, Hypertrophic | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- B-Cell Acute Lymphoblastic Leukemia/Diffuse Large B-Cell Lym (Experimental): Participants will have relapsed or refractory B-Cell Acute Lymphoblastic Leukemia or Diffused Large B-Cell Lymphoma
  Interventions: Drug: 131-I Apamistamab; Biological: CAR T-cell

INTERVENTIONS:
Drug: 131-I Apamistamab — Patients will receive 131-I apamistamab 5-7 days prior to a single infusion of 1x10^6 19-28z CAR T-cells/kg for those in the B-ALL cohort, or 2x10^6 19-28z CAR T-cells/kg, for those in the DLBCL. 131-I apamistamab may be administered inpatient or outpatient at the discretion and judgment of the treating investigators.
  Other Names: Iomab-B
Biological: CAR T-cell — 19-28z CAR T-cells will be administered inpatient as a single infusion of 1x10^6 19-28z CAR T-cells/kg, for those in the B-ALL cohort, or 2x10^6 19-28z CAR T-cells/kg, for those in the DLBCL cohort. Patients will be observed inpatient for a minimum of 7 days (longer as clinically indicated and at the discretion of the treating physician).

SUMMARY:
This is a pilot study; patients will receive 131-I apamistamab prior to CAR T-cell infusion in order to determine the maximum tolerated dose of 131-I apamistamab is exceeded at 75 mCi, and if so, to assess the safety of a step-down dose of 50 mCi.

ELIGIBILITY:
Patients with B-ALL or DLBCL (or subtypes thereof) who have relapsed or refractory disease will be eligible. Refractory disease is defined by failure to achieve at least a partial response or disease progression within 6 months of the last therapy. Patients who initially respond but subsequently demonstrate disease progression are considered to have relapsed disease

Participant Inclusion Criteria:

- To be eligible for leukapheresis, patients must have a CD19+ B-cell malignancy with relapsed or refractory disease, defined below. To be eligible for 131-I apamistamab conditioning and treatment with 19-28z CAR T-cells, patients must additionally have detectable evidence of residual malignancy at the time of assessment prior to CAR T-cell infusion (as defined below), regardless of therapy administered following leukapheresis.

a. Patients with diffuse large B-cell lymphoma (de novo or DLBCL transformed from an indolent lymphoma (follicular lymphoma, chronic lymphocytic leukemia [Richter syndrome]) or high-grade B-cell lymphoma (HGBL): ("DLBCL patients") i. Defined as relapsed or refractory DLBCL or high-grade B-cell lymphoma (HGBL) following 2 or more prior chemoimmunotherapy regimens (with at least one course including an anthracycline and CD20-directed therapy) following diagnosis of de novo DLBCL/HGBL or DLBCL arising from indolent lymphoma, and requiring further treatment. Exception: patients with Richter syndrome (DLBCL arising from CLL/small lymphocytic lymphoma) are eligible following 1 or more prior chemoimmunotherapy regimens (with at least one course including an anthracycline and CD20-directed therapy) and do not require a second course of chemoimmunotherapy to be eligible.

ii. Patients must have at least one FDG-avid (PET-avid) measurable lesion iii. Biopsy confirmation of relapsed of refractory DLBCL is required iv. For patients who have received treatment for confirmed relapsed or refractory disease otherwise meeting criteria a.i.-a.iii. as above, within 6 weeks of study enrollment, active disease does not need to be re-confirmed or present immediately prior to Screening A for the patient to be eligible for leukapheresis. However, detectable evidence of residual malignancy must be present at Screening B in order for the patient to be eligible for 131-I apamistamab and CAR T-cell therapy.

b. Patients with B-cell acute lymphoblastic leukemia or B lymphoblastic lymphoma (ALL) or chronic myeloid leukemia (CML) in lymphoid blast crisis: ("B-ALL patients") i. Patients with Philadelphia chromosome-negative B-cell ALL must have been refractory to at least 1 line of multi-agent chemotherapy or relapsed following at least 1 prior multiagent systemic chemotherapy regimen that included induction and consolidation therapy ii. Patients with Philadelphia chromosome-positive ALL or CML in lymphoid blast crisis must have exhibited persistent disease following therapy with a second- or third-generation tyrosine kinase inhibitor iii. Patients must have ≥5% bone marrow involvement and/or at least one FDG-avid (PET-avid) measurable extramedullary lesion iv. For patients who have received treatment for confirmed relapsed or refractory disease otherwise meeting criteria b.i.-b.iii. as above, within 6 weeks of study enrollment, active disease does not need to be re-confirmed or present immediately prior to Screening A for the patient to be eligible for leukapheresis. However, detectable evidence of residual malignancy must be present at Screening B in order for the patient to be eligible for 131-I apamistamab and CAR T-cell therapy.

* While prior CD19-targeted therapies, including CAR T-cell therapy, do not exclude participation, CD19 expression by immunohistochemical staining or flow cytometry must be confirmed prior to enrollment.
* Age ≥ 18 years of age
* Creatinine clearance ≥50 mL/min as calculated by the Cockroft-Gault formula
* Direct bilirubin ≤2.0 mg/dL, AST and ALT ≤3.0x upper limit of normal (ULN), unless liver dysfunction is thought to be related to underlying malignancy
* Adequate pulmonary function as assessed by ≥92% oxygen saturation on room air by pulse oximetry.
* Adequate bone marrow function meeting the following criteria as defined below, without requiring blood product or granulocyte-colony stimulating factor support in the past 7 days, unless cytopenias are attributed to underlying malignancy in the opinion of the investigator:

  1. Absolute neutrophil count ≥0.5k/µL,
  2. Platelets ≥30k/µL,
  3. Hemoglobin ≥7g/dL.
* ECOG performance status 0-2.

Participant Exclusion Criteria:

* ECOG performance status ≥3.
* Pregnant or lactating patients. Patients of childbearing age should use effective contraception while on this study and continue for 1 year after all treatment is finished.
* Impaired cardiac function (LVEF <40%) as assessed by echocardiogram or MUGA scan during screening
* Patients with active graft versus host disease following allogeneic hematopoietic cell transplantation requiring systemic T-cell suppressive therapy are ineligible
* Patients with active autoimmune disease requiring systemic T-cell suppressive therapy are ineligible
* Patients with following cardiac conditions will be excluded:

  1. New York Heart Association (NYHA) stage III or IV congestive heart failure
  2. Myocardial infarction ≤6 months prior to enrollment
  3. Any history of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration
  4. Any history of severe non-ischemic cardiomyopathy with LVEF ≤20%
* Have current or prior positive test results for human immunodeficiency virus (HIV) or hepatitis B (HBV) or C (HCV), with the following exceptions:

  1. Subjects who have positive HBV test results due to having been previously vaccinated against hepatitis B, as evidenced by negative hepatitis B surface antigen (HBsAg), negative anti- hepatitis B core protein (HBc) and positive antibody to the HBsAg (anti-HBs) are not excluded.
  2. Subjects who have antibodies to HCV or who have hepatitis B core antibody, with undetectable viremia by PCR, and with adequate organ function as defined in the protocol, are not excluded.
* Patients with uncontrolled systemic fungal, bacterial, viral or other infection are ineligible.
* Patients with any concurrent active malignancies as defined by malignancies requiring any therapy other than expectant observation or hormonal therapy, with the exception of squamous and basal cell carcinoma of skin.
* Patients with history or presence of clinically significant neurological disorders such as epilepsy, generalized seizure disorder, severe brain injuries are ineligible.
* Any other issue which, in the opinion of the treating physician, would make the patient ineligible for the study.
* Patients with circulating human anti-mouse antibodies to BC8 noted on initial screening (see Appendix III)

Subject Inclusion Criteria for 131-I Apamistamab Infusion Patients should meet performance status and organ function parameters as specified, without known development of an exclusion criterion, prior to proceeding to 131-I apamistamab infusion. See Section 9.2 re: screening for treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-02-02 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities and maximum tolerated dose of 131-I apamistamab, when given in combination with 19-28z CAR T-cells for treatment of relapsed or refractory B-cell ALL or DLBCL | 30 days after treatment
  To determine the safety and tolerability of a single dose of 131-I apamistamab given prior to 19-28z CAR T-cell infusion in patients with relapsed or refractory B-cell ALL or DLBCL.

CONTACTS AND LOCATIONS:
Overall Officials: Mark B Geyer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org